CLINICAL TRIAL: NCT02423213
Title: Determination of Feasibility of Intraoperative Spectral Domain Microscope Combined/Integrated OCT Visualization During En Face Retinal and Ophthalmic Surgery: DISCOVER Study
Brief Title: DISCOVER Study: Microscope-integrated Intraoperative OCT Study
Acronym: DISCOVER
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Justis Ehlers, Assistant Professor of Ophthalmology, The Cleveland Clinic
Other Study IDs: 14-013; K23EY022947-01A1 (NIH)
Record Dates: First submitted 2015-04-08; First posted 2015-04-22 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Retinal Diseases; Fuchs Endothelial Dystrophy; Macular Hole; Epiretinal Membrane; Retinal Detachment
Keywords: OCT; image-guided surgery; ophthalmic surgery
MeSH Terms: conditions — Retinal Diseases; Fuchs' Endothelial Dystrophy; Retinal Perforations; Epiretinal Membrane; Retinal Detachment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Optical coherence tomography (OCT )provides high resolution information regarding the anatomic structure of the tissues of the eye in a cross-sectional and 3 dimensional view. Much of this information is not able to be visualized by a clinician. Utilizing this information during surgery will allow for the ophthalmic surgeons to better understand how surgical procedures impact the anatomic structure of the eye.

In this study an OCT device that has been built into the microscope (rather than mounted on the side or held in the surgeon's hand) and will be utilized to take images at various milestones during surgery to assess feasibility and potential utility of this technology. Since it is built into the microscope, there are potential significant advantages over a separate system including increased efficiency, improved working distance, and the ability to visualize tissue-instrument interactions.

DETAILED DESCRIPTION:
Optical coherence tomography (OCT) has become a critical component to the evaluation of ophthalmic disease. Similar to the ultrasound, OCT uses light to reconstruct an image of the tissue of interest. In effect, OCT functions almost like a light biopsy, allowing clinicians to visualize subtle changes in the tissue, such as macular edema or subretinal fluid. OCT in the clinic setting has become the gold standard for monitoring diseases such as macular degeneration and diabetic retinopathy;and it has become one of the most frequently ordered diagnostic test in ophthalmology.

Due to the restraints in the size and structure of the imaging equipment, the use of OCT in the operating room has been limited. More recently, modifications to OCT table-tops models as well as the development of hand-held OCT probes have allowed for the translation of OCT technology into the operating room. The high resolution anatomic information that is gained from the OCT imaging is a natural complement to the ophthalmic surgeon. Using OCT during vitreoretinal surgery has revealed subtle changes in the microarchitecture of the retinal diseases such as retinal detachment, macular hole and optic pit, that were not previously known. Our research team has been examining intraoperative OCT in the operating room using both a handheld and microscope-mounted portable spectral domain OCT probe with excellent success and an outstanding safety record.

In this study an OCT device that has been built into the microscope (rather than mounted on the side or held in the surgeon's hand) and will be utilized to take images at various milestones during surgery to assess feasibility and potential utility of this technology. Since it is built into the microscope, there are potential significant advantages over a separate system including increased efficiency, improved working distance, and the ability to visualize tissue-instrument interactions.

ELIGIBILITY:
Inclusion Criteria:

* The study population includes any patient requiring ophthalmic surgery

Exclusion Criteria:

* Under the age of 18 years.
* Cognitive/Mentally impaired or unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes any patient requiring ophthalmic surgery who meets the inclusion criteria for feasibility of OCT imaging.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To assess feasibility of microscope-integrated intraoperative OCT | 3 years
  Feasibility will be assessed as the percentage of cases where OCT images were successfully obtained with a microscope-integrated system

SECONDARY OUTCOMES:
To assess utility of microscope-integrated intraoperative OCT on surgical decision-making | 3 years
  Utility will be assessed through a surgeon-feedback questionnaire, including the percentage of cases where the OCT information changed the surgical approach to the case according to the surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Justis P Ehlers, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehlers JP, Srivastava SK, Feiler D, Noonan AI, Rollins AM, Tao YK. Integrative advances for OCT-guided ophthalmic surgery and intraoperative OCT: microscope integration, surgical instrumentation, and heads-up display surgeon feedback. PLoS One. 2014 Aug 20;9(8):e105224. doi: 10.1371/journal.pone.0105224. eCollection 2014. PMID 25141340
- [Background] Ehlers JP, Kaiser PK, Srivastava SK. Intraoperative optical coherence tomography using the RESCAN 700: preliminary results from the DISCOVER study. Br J Ophthalmol. 2014 Oct;98(10):1329-32. doi: 10.1136/bjophthalmol-2014-305294. Epub 2014 Apr 29. PMID 24782469